CLINICAL TRIAL: NCT03898622
Title: Supplementation of Thyroid Hormone for TSH Control in Patients With Chronic Kidney Disease Without Renal Replacement Therapy: Randomized, Double-blind Clinical Trial at Guadalajara Civil Hospital.
Brief Title: Supplementation of Thyroid Hormone for TSH Control in Patients With Chronic Kidney Disease Without TRR.
Acronym: TSHrenal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Guillermo Navarro Blackaller, resident of nephrology, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HospitalCG 034/18
Record Dates: First submitted 2018-08-28; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Diseases; Subclinical Hypothyroidism
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: Phase II study, type placebo controlled clinical trial, randomized of two arms, double blind, unicentric.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study drug and placebo will be packaged and labeled on the basis of this randomization program, being letters both, for placebo or Levothyroxine, coding that only the third randomization investigator outside the study will know. The letters of the drugs will be preprinted on the study drug labels and will be assigned to double blind treatment as the subjects meet the requirements for the study Both groups treated with fasting medication (levothyroxine) (in the case of taking a drug that interacts with absorption, use of the drug is changed according to the specified hours, see Table 2) or fasting placebo according to the randomization 1: 1 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with levothyroxine (Active Comparator): Patients with Chronic Kidney Disease G2-G5 with proteinuria without renal replacement therapy, who comes to the clinic of renal health clinic of Fray Antonio Alcalde civil hospital. That meet the inclusion criteria. Levothyroxine 25 mcg (1/4 tablet of 100mcg) was administered in fasting the first month, the doctor evaluated with monthly control of TSH levels (if the TSH level was not in the range of TSH 1-2.5 uim / L the second month increase to a dose of 50 mcg (1/2 tablet of 100mcg fasting, or similarly if the patient had a TSH <1 u / L was suspended in medication and it was valued restart the next month the medication if TSH> 2.5u / L ) to complete three months of intervention.
  Interventions: Drug: Levothyroxine
- Group Placebo (Placebo Comparator): atients with Chronic Kidney Disease G2-G5 with proteinuria without renal replacement therapy, who comes to the clinic of renal health clinic of Fray Antonio Alcalde civil hospital. that meet the inclusion criteria.
  Placebo (1/4 tablet) was administered in fasting the first month, the doctor assessed with monthly control of TSH levels (if the TSH level was not in the range of TSH 1-2.5 UM / L the second month increase at a dose (1/2 tablet fasting, or similarly if the patient had TSH <1 u / L was suspended in medication and it was valued restart the next month the medication if TSH> 2.5 / month) to complete three months of intervention.
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — levothyroxine with a safe dose for our population with high cardiovascular risk of 0.25mcg so that the patient's weight range between 50-80kg maintains a dosage of 0.3-0.5mcg / kg / day that does not affect the thyroid axis) fasting levothyroxine (in the case of taking a drug that interacts with absorption, use of it is changed according to the specified hours, see Table 2), and adjusted according to TSH levels > 1 and normal T4L
  Other Names: placebo

SUMMARY:
Study design: Phase II study, randomized, double-blind, unicentric, two-arm, placebo-controlled clinical trial. Methods and participants: Patients with Chronic Kidney Disease G2-G5 with proteinuria without renal replacement therapy, who come to the clinic of renal health clinic of the Fray Antonio Alcalde civil hospital. As criteria for non-inclusion, need for dialysis, primary hypothyroidism or pre-existing thyroid disease, ischemic heart disease in a period less than 6 months, arrhythmia, pregnancy, use of drugs that interact with synthesis of thyroid hormones, do not accept informed consent, thyroid stimulating hormone (TSH) <2.5 uiml / L or TSH> 10 uiml / L.

DETAILED DESCRIPTION:
Thyroid disorders, especially elevated TSH levels in patients with CKD, are frequent. As it is an easy medication to acquire and of little cost compared to the other options, levothyroxine would provide benefits already known in patients with CKD and also a proteinuria effect (knowing each other). as a factor of progression of the CKD a health problem worldwide) being a potentially useful treatment and a dose that the risk is minimal. The study consists of 3 phases, the first phase consists of capturing patients from the renal health clinic, having baseline measurement of the variables. Then, the second phase consists of both groups treating them with medication (levothyroxine with a safe dose for the investigator's population with high cardiovascular risk of 0.25mcg so that the patient's weight range between 50-80kg maintains a dosage of 0.3-0.5mcg / kg / day that the thyroid axis is not affected) of fasting levothyroxine (in the case of taking a drug that interacts with absorption changes its use according to the specified hours, see Table 2) or placebo according to the randomization 1: 1 for three months and that have treatment with ACEI or ARA-2 (specifying which and the dose thereof), with follow-up every 4 weeks (Monitoring thyroid function). The third phase consists of a comparison of the variables studied.

The primary objective is to evaluate the effect of the use of levothyroxine on the levels of proteinuria measured on the test strip of the general urine and protein examination in 24-hour urine patients with chronic kidney disease without renal support therapy with proteinuria, who already receive the standard antiproteinuric treatment with an ACE inhibitor or ARA-2 against placebo and the secondary objectives are to evaluate the changes in proteinuria, according to TSH levels in 2.5-9.9 μiml /L, with the levels of T4L in levels 0.8-1.8mcg / ml), analyze improvement in glomerular filtration rate in patients receiving levothyroxine and at the end of the study and evaluate Tolerability and safety of levothyroxine as antiproteinuric treatment in chronic kidney disease without renal support therapy, and as secondary objectives improvement in cholesterol, triglycerides blood pressure. Any adverse event will be recorded in the adverse event reporting forms. (definition of the International Conference on Harmonization [ICH])

ELIGIBILITY:
Inclusion Criteria:

* • Patients older than 18 years

  * Patients with chronic kidney disease G2-G5 without renal replacement therapy) who attend a renal health clinic.
  * Presence of proteinuria in a test strip, 24 hours urine collection (greater than 150mg / dl in 24hrs urine)
  * TSH <9.9uiml / L and TSH> 2.4 0uiml / L
  * Take an IECA or ARA-2
  * Patients with weight> 50 kg and <80kg
  * Accept informed consent

Exclusion Criteria:

* Chronic dialysis (peritoneal dialysis or hemodialysis)

  * Primary hypothyroidism or preexisting thyroid disease
  * Use of levothyroxine.
  * TSH> 10uiml / L and TSH <2.5 0uiml / L
  * Positive thyroid antibodies
  * Ischemic heart disease in less than 6 months
  * Cardiac arrhythmia
  * Use Medications (Levothyroxine synthesis, see Table 2)
  * Anxiety disorder
  * Pregnancy
  * Do not accept consent
  * Patients weighing <50 kg and> 80kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
24 hours urine Proteinuria in patients with subclinical hypothyroidism and CKD G2-G5 without renal support therapy Randomized clinical trial of levothyroxine group versus placebo | three months
  24 hours urine Proteinuria in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy, in two study arms the first in patients with the use of levothyroxine in 18 patients (TSH in a safe range 1-2.5 μm / L ), in patients who already use ACE inhibitors or ARA-2 (at least 3 months), versus the second arm in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy in patients who already use ACE inhibitors or ARA- 2 (at least 3 months) with placebo in 14 patients, Based on proteins in 24-hour urine collection at the beginning and end of three months. with follow-up every 4 weeks (Monitoring thyroid function and adjusting dose in a safe range TSH 1-2.5uim / L).

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) in patients with subclinical hypothyroidism and CKD G2-G5 without renal support therapy Randomized clinical trial of levothyroxine group versus placebo | three months
  Estimated glomerular filtration rate in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy, in two study arms the first in patients with the use of levothyroxine in 18 patients (TSH in a safe range 1-2.5 μm / L), versus the second arm in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy with placebo in 14 patients, Based on the measurement of creatinine serica (MDRD formula was used to calculate eGFR expressed in ml/min/1.73m2) at the beginning and end of three months. with follow-up every 4 weeks (Monitoring thyroid function and adjusting dose in a safe range TSH 1-2.5uim / L).
Measurement of lipid profile (cholesterol, LDL and triglycerides) in patients with subclinical hypothyroidism and CKD G2-G5 without renal support therapy Randomized clinical trial of levothyroxine group versus placebo. | three months
  Measurement of lipid profile (Cholesterol, LDL cholesterol and triglycerides) in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy, in two studies in the patients with the use of levothyroxine in 18 patients (TSH in a safe range 1-2.5 μm / L), versus the second arm in patients with subclinical hypothyroidism and chronic kidney disease G2-G5 without renal support therapy with placebo in 14 patients, Based on the measurement of cholesterol, triglycerides and serum LDL expressed in mg / dl at the beginning and end of three months. with follow-up every 4 weeks (Monitoring thyroid function and adjusting dose in a safe range TSH 1-2.5uim / L).

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) when using levothyroxine in patients with subclinical hypothyroidism and CKD | four months
  with follow-up every 4 weeks, with thyroid profile control tests and adverse effects will be reported and follow-up. It will be valued in accordance with intensity According to the criteria CTC v. 3.0 (1-5), start date and end thereof, as well as the treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chavez, Study Director — Hospital Civil de Guadalajara
Locations (1):
- Kidney health clinic, Civil Hospital of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT03898622/Prot_SAP_ICF_000.pdf